CLINICAL TRIAL: NCT04934488
Title: Online 1-Day Peer-Delivered Cognitive Behavioural Therapy (CBT)-Based Workshops for Postpartum Depression
Brief Title: Online Peer-Delivered 1-Day CBT Workshops for PPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Ryan Van Lieshout, MD, PhD, Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Peer1DayCBT
Record Dates: First submitted 2021-05-13; First posted 2021-06-22 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): The experimental (immediate workshop) group will receive the online workshop at baseline (T1). The experimental group will also receive care as usual from their healthcare providers.
  Interventions: Behavioral: Online Peer-Delivered 1-Day CBT-Based Workshop
- Waitlist Control (Other): The waitlist control group will receive care from usual healthcare providers and will receive the intervention at the conclusion of the study period (T2, 12 weeks after enrollment).
  Interventions: Behavioral: Online Peer-Delivered 1-Day CBT-Based Workshop

INTERVENTIONS:
Behavioral: Online Peer-Delivered 1-Day CBT-Based Workshop — It is a day-long intervention delivered in 4 modules. Each participant is given a professionally designed manual to facilitate learning. The 1st contains information on PPD etiology with a focus on modifiable cognitive risk factors (e.g., negative thoughts, maladaptive core beliefs). The 2nd module focuses on cognitive skills including cognitive restructuring. The 3rd builds behavioural skills such as problem solving, behavioural activation, assertiveness, sleep strategies, and using supports. The final module provides an opportunity for goal setting/action planning. Teaching methods include didactic sections, group exercises, and role-plays.

SUMMARY:
A parallel group RCT with experimental (immediate workshop) and waitlist control (treatment 12 weeks later) groups will address our objectives. All participants will be asked to complete study questionnaires at baseline (T1, 3 weeks before the intervention/first workshop) and 12 weeks later (T2, just prior to the waitlist control/second workshop). Workshops will be delivered by trained peer leaders (women who have recovered from PPD). The study will aim to determine if online 1-day CBT-based workshops for PPD delivered by trained lay peers added to care as usual during the COVID-19 pandemic: (1) can improve PPD more than usual care alone, (2) are cost-effective, (3) can reduce the impact of common comorbidities and complications of PPD including anxiety, partner-relationship discord, social support, infant temperament, parenting stress, and poorer mother-infant attachment.

DETAILED DESCRIPTION:
The COVID-19 pandemic has further exposed vulnerabilities in social and economic systems that lead to inequalities for mothers with mental health problems and their children, worsening unintended systematic biases that exist within the healthcare system. Women with postpartum depression (PPD) are experiencing substantial worry (1), isolation, loneliness, and insomnia (2), all of which have increased levels of PPD(3,4). Mothers now have more responsibilities than ever before, providing care to their infants and toddlers, educating their older children, managing households, and supporting their partners. They are also profoundly worried about job losses, reduced income, and food insecurity (5), all of which have disrupted family routines and increased levels of partner conflict and rates of intimate partner violence.(6)

Postpartum depression (PPD) typically affects up to 1 in 5 women (7-9) and increases the risk of later depressive episodes (10), parenting problems (11), poor mother-infant attachment (12), and emotional, behavioural, and school problems in offspring (13,14). A single case of PPD has been estimated to cost as much as $150,000 over the lifespan (15), or $57 billion for each annual cohort of Canadian births.

Even under ideal conditions, the healthcare system is poorly equipped to provide care for problems requiring urgent psychotherapy like PPD (e.g., just 1 in 10 women with PPD receive evidence-based care) (16). Barriers include women's preference for psychotherapy over medication, a lack of time, and a reluctance to travel to regular appointments (17,18). During the pandemic, the healthcare system has become even less able to help these women as public health units that previously supported the mental health of mothers have shifted their priorities to direct COVID response. Moreover, social distancing recommendations aimed at reducing COVID-19 risk have inadvertently increased psychological distress (19) and decreased access to resources that protect against PPD including social and practical support from family, friends, and professionals.

Peer administered interventions (PAIs - those delivered by recovered former patients) are increasingly recognized as potentially effective alternatives to traditional mental health care services (21). Such treatments capitalize on the fact that in the case of psychotherapy, it is not clear that the level of training predicts treatment quality or outcome (22,23) for patients. Depression is an appropriate target for PAIs because it is relatively common, there is substantial unmet treatment need, and recovery rates are high, suggesting that peers will be widely available (21). The few studies that have examined the impact of PAIs for depression suggest they can be effective in both the short and long term but are most effective if: a) they are delivered by peers alone, and b) structured and based on evidence-based treatments (rather than providing non-specific support) (21). In the context of the COVID-19 pandemic peer-delivered interventions are particularly appealing, considering redeployment and re-prioritizing of healthcare providers and services to focus on responding to the pandemic.

Only interventions that are considered safe and that can be rapidly upscaled can have an impact on PPD at the population level (24). Ideal large-scale interventions for PPD during the COVID-19 pandemic are not only safe (i.e., delivered online), but brief, utilize the treatments most preferred by women (i.e., non-pharmacological), reduce barriers to accessibility (i.e., self-referred), provide skills that can be used over the long-term, and delivered in large groups to increase social support. At present time, no interventions exist that meet all of these criteria.

Research Questions Primary Research Question: Can Online 1-Day CBT-Based Workshops for PPD delivered by trained lay peers added to care as usual during the COVID-19 pandemic improve PPD more than usual care alone? Secondary Research Question: Are the workshops cost-effective? Tertiary Research Question: Can these workshops reduce the impact of the common comorbidities and complications of PPD (anxiety, partner relationship discord, social support, infant temperament, parenting stress, and poorer mother-infant attachment)?

Design A parallel group RCT with experimental (immediate workshop) and waitlist control (treatment 12 weeks later) groups will address our objectives. All participants will be asked to complete study questionnaires at baseline (T1, 3 weeks before the intervention/first workshop) and 12 weeks later (T2, just prior to the waitlist control/second workshop). Peers delivering groups will be randomly assigned to workshops and not notified of group status.

Intervention: The experimental (immediate workshop) group will receive the online workshop at baseline (T1), and the control (waitlist) group will receive the intervention twelve weeks later. Both groups can also receive care as usual from their healthcare providers.

The online workshop was developed by the NPI, Ryan Van Lieshout (a perinatal psychiatrist who has developed and tested effective brief group CBT for PPD interventions), Peter Bieling (author of the world's leading group CBT manual), and June Brown (developer of 1-Day CBT-Based workshops for depression in the UK). It is a day-long intervention delivered in 4 modules. Each participant is given a professionally designed manual (Attached) to facilitate learning. Weekly reminder emails are sent for 8 weeks after workshop completion to encourage practice. The investigators also provide a list of PPD resources and a copy of the Canadian Practice Guidelines for the Treatment of PPD (written by NPI).

Lay peers who have recovered from PPD will be recruited (n=5) to be trained to deliver the workshops. The investigators will utilize the CBT training program and screening and safety protocols (e.g., handling suicidality, child safety issues) developed in the context of a previous study where a psychologist and psychotherapist delivered the 1-Day CBT workshops.

Given the situation with COVID-19, the investigators will run the CBT workshops virtually via ZOOM.

Randomization: Women will undergo block randomization to the experimental or waitlist control group using permuted block sizes of 4, 6, and 8. The randomization scheme will be generated in the statistical computing program R. The randomization of participants will be delivered to the research coordinator via the online REDCap (Research Electronic Data Capture) system. The investigators will track reasons for loss to follow-up.

Recruitment: The investigators will recruit participants via social and online media, our public health and community partners, midwifery groups, and obstetrical and family practices.

ELIGIBILITY:
Inclusion Criteria:

* reside in Ontario
* have an infant <12 months old
* 18 years or older
* EPDS score 10 or more

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Depression | 12 weeks
  The Edinburgh Postnatal Depression Scale (EPDS) is the 10-item gold standard measure of PPD. Total scores range from 0-30 with higher scores indicating worse depressive symptoms.. A score ≥13 is consistent with PPD and changes in scores >4 are accepted as being indicative of clinically significant change (31).

SECONDARY OUTCOMES:
Cost-Effectiveness - Costs | 12 weeks
  Cost-effectiveness will be measured using incremental cost per quality-adjusted life year ratio.
  Costs: Healthcare resource utilization data (including mental health service use) will be collected using a questionnaire based on the Canadian Community Health Survey and the Service Use and Resources Form, adapted for the postpartum period and used in previous PPD research. Corresponding unit costs will be calculated using provincial or other standard billing rates.
Cost-Effectiveness - Quality Adjusted Life Year | 12 weeks
  Cost-effectiveness will be measured using incremental cost per quality-adjusted life year ratio.
  Quality-Adjusted Life Year (QALY): The EQ-5D-5L is a utility-based health-related quality of life instrument consisting of five questions covering depression/anxiety, usual activities, self-care, pain/ discomfort, and mobility. For each participant, a QALY will be calculated by multiplying the health utility for the matching time period (i.e., the area under the curve approach).
Anxiety | 12 weeks
  The Generalized Anxiety Disorder 7-Item Scale (GAD-7) (32) is a self-report scale that taps generalized anxiety disorder, the most common comorbidity of PPD. Items are scored on a 4-point scale from 0 to 3, with a higher score indicating an increased risk of GAD. The GAD-7 will be examined as both a continuous and dichotomous outcome, where a cutoff of ≥11 defined clinically important levels of anxiety symptoms.
Mother-Infant Bonding | 12 weeks
  Postpartum Bonding Questionnaire (PBQ) is a 25-item measure that will be used to assess 3 aspects of maternal-infant relations: (1) bonding, (2) rejection and anger towards the infant, (3) infant-focused anxiety. Each item is scored on a scale of 0-5, with higher scores suggestive of more problems. Mother-infant bonding will be measured as a continuous and dichotomous outcome, using cut-off scores for each subscale indicating bonding disorders. Cutoff values of 12 for the bonding subscale, 17 for rejection and anger, and 10 for infant-focused anxiety have been proposed to define bonding disorders in each category.
Social Support | 12 weeks
  The Social Provisions Scale (SPS) is a 24-item self-report measure of the degree to which the social relationships within an individual's life provide support. Items are scored on a 4-point scale (1-4) and total scores range from 24-96, with higher scores indicating more perceived support.
Partner Relationship Quality | 12 weeks
  The Dyadic Adjustment Scale is a 32-item questionnaire that measures an individual's perceptions of his/her relationship with an intimate partner. Questions are answered on 6-point scales. Totals cores vary from 0-151 with higher scores indicating better perceived dyadic relationship.
Parenting stress | 12 weeks
  The Parenting Stress Index (short form) is a 36-item parent self-report measure that identifies potentially dysfunctional parent-child systems on three subscales: parental distress, parent-child dysfunctional interaction, and difficult child. The measure also produces a total score that is an indication of overall level of stress a person is feeling in their role as a parent. Higher scores indicate higher levels of stress.
Infant Temperament | 12 weeks
  The Infant Behaviour Questionnaire-Revised (Very Short Form) (IBQR) is a parent-report measure of infant temperament. The IBQ-R (Very Short Form) consists of 37 items answered on a 7-point scale (1-7) and assesses 3 factors: Positive Affectivity/Surgency with 13 items, Negative Emotionality with 12 items, and Orienting/Regulatory Capacity with 12 items; higher scores indicate greater alignment with the domain.
Client Satisfaction | 12 weeks
  Satisfaction with the workshop will be assessed using the CSQ-8, an 8-item self-report scale. Items are scored using a 4-point likert-scale with total scores ranging from 8-32. Higher scores indicated higher satisfaction. The CSQ-8 will be analyzed using the continuous scale score for participants who complete the intervention in the experimental arm of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Van Lieshout, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Drage JT, Layton H, Varambally M, Jack SM, Van Lieshout RJ. Birthing parents' perceptions of an online peer-delivered 1-day cognitive-behavioural therapy-based workshop for postpartum depression added to usual care. Midwifery. 2025 Apr;143:104319. doi: 10.1016/j.midw.2025.104319. Epub 2025 Jan 30. PMID 39923292